CLINICAL TRIAL: NCT06803810
Title: Peer to Peer (P2P): Mental Health Interventions With Persons With Substance Use Disorders
Acronym: P2P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: South Carolina Center for Rural and Primary Healthcare (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2220242
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Standard of Care; P2P Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): This group will complete a baseline, week 6, and week 12 study visit. Participants will complete research visits (in-person or virtually) at which time they will complete a series of questionnaires.
- P2P Intervention (Experimental): This group will complete the same study visits as the standard care group with an additional week 3 visit and 6 CPSS-led therapy intervention sessions. These CPSS led sessions will be completed by the end of the 12week study period. At each study visit you will complete questionnaires.
  Interventions: Behavioral: P2P Intervention

INTERVENTIONS:
Behavioral: P2P Intervention — This group will complete the same study visits as the standard care group with an additional week 3 visit and 6 CPSS-led therapy intervention sessions. These CPSS led sessions will be completed by the end of the 12week study period. At each study visit you will complete questionnaires.
  Arms: P2P Intervention

SUMMARY:
This study provides substance use and mental health peer support services to address behavioral health disparities in rural areas. Specifically, the project aims to address persistent mental health symptoms, such as anxiety and depression, that become barriers to care for patients working towards long-term recovery from co-occurring mental health and substance use disorders. Participants will be assessed and evaluated for opioid use disorder (OUD), social determinants of health (SDoH), and infectious diseases by a nurse practitioner and a social worker. A certified peer support specialist (CPSS) will provide additional support, connecting patients to sustainable mental health resources and implementing a modified version of the Friendship Bench intervention, which involves six weekly 45-minute problem-solving therapy sessions with the option to participate in six or more peer support sessions. The CPSS will follow the patient for up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OUD via Diagnostic Statistical Manual (DSM)-V Text Revision (TR)
* Receiving MOUD through the Mobile Recovery Program for at least 3 months
* Age 18 or older
* Moderate to Severe Depression with or without co-occurring anxiety as determined by PHQ-9 conducted during the most recent MRP clinical visit

Exclusion Criteria:

* Severe cognitive, medical, or psychiatric disability that could impair ability to perform study-related activities as determined by the MRP clinician or principal investigator.
* Unable to read/speak English
* Unable to read and comprehend the consent materials and other study materials
* Current suicidal ideation based on the Patient Health Questionnaire-9

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-12-29 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
Reduction in depressive symptoms | 12 weeks
  Reduce depression symptoms as measured by the PHQ-9

CONTACTS AND LOCATIONS:
Overall Officials: Alain Litwin, Principal Investigator — Prisma Health
Locations (1):
- Prisma Health, Greenville, South Carolina, United States